CLINICAL TRIAL: NCT01442285
Title: The Mental Health and Dynamic Referral for Oncology Protocol (MHADRO)
Acronym: MHADRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Polaris Health Directions (Industry)
Responsible Party: Principal Investigator, Edwin Boudreaux, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MHADRO; H-13561 (Other: UMass IRB); R42MH078432 (NIH)
Record Dates: First submitted 2011-04-16; First posted 2011-09-28 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Cancer; Distress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- personalized, motivational messages (Experimental): A Healthcare Provider Report will be reviewed by oncologist. If mental health functioning scores are elevated or high range,treatment plan is constructed. Subjects receive personalized Patient Feedback Report after each assessment which will include motivationally tailored messages and suggestions for action.
  Interventions: Behavioral: personalized, motivational messages
- Control Group (No Intervention): Control subjects will receive a resource packet upon initial diagnosis consisting of brochures and printed material describing local resources and support groups as part of their routine care. At 12 months, subjects will receive the full assessment with reports and referrals.

INTERVENTIONS:
Behavioral: personalized, motivational messages — A Healthcare Provider Report will be printed after each assessment and reviewed by the subject's oncologist. If any mental health functioning scale scores fall in the elevated or high range, a treatment plan will be constructed. Subjects will receive a personalized Patient Feedback Report after each assessment which will include motivationally tailored messages and suggestions for action.
  Other Names: motivational counseling
  Arms: personalized, motivational messages

SUMMARY:
The purpose of this study is to understand more about meeting the psychosocial needs of people who have cancer.

DETAILED DESCRIPTION:
The investigators are interested in the feasibility of using computer assisted screening and assessment to meet the psychosocial needs of people with cancer. The investigators are studying two different interventions. Both groups will receive health information, referral information, and resources. One group will also receive tailored feedback reports.

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Decrease in psychological stress | 12 months
  Both groups will receive a full assessment, referral information, and resources. Only the intervention group will have the option of immediately sending their contact information to a counselor/mental health provider and receive a tailored feedback report with specific recommendations about managing their psychological and social needs, and provide education about ways to improve their quality of life. We anticipate that distressed subjects assigned to the Intervention Group will exhibit larger decreases in psychological distress when compared against the Control Group.

SECONDARY OUTCOMES:
Reduced distress | 12 months
  Reduced distress will be achieved through initiation of mental health counseling, psychotropic medications, and psychosocial support group participation in distressed patients who are not currently receiving mental health treatment at baseline, and enhancement of existing mental health treatment in patients already receiving some form of mental health treatment at baseline, including adding another treatment modality, such as psychotherapy being added to a medication regimen, or adjusting their existing mental health treatments, such as increasing the dose of an anti-depressant.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Boudreaux, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, UMass Memorial, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] O'Hea E, Kroll-Desrosiers A, Cutillo AS, Michalak HR, Barton BA, Harralson T, Carmack C, McMahon C, Boudreaux ED. Impact of the mental health and dynamic referral for oncology (MHADRO) program on oncology patient outcomes, health care utilization, and health provider behaviors: A multi-site randomized control trial. Patient Educ Couns. 2020 Mar;103(3):607-616. doi: 10.1016/j.pec.2019.10.006. Epub 2019 Nov 5. PMID 31753521
- [Derived] O'Hea EL, Monahan BR, Cutillo A, Person SD, Grissom G, Boudreaux ED. Predictors of psychological distress and interest in mental health services in individuals with cancer. J Health Psychol. 2016 Jun;21(6):1145-56. doi: 10.1177/1359105314547752. Epub 2014 Sep 9. PMID 25205777